CLINICAL TRIAL: NCT03543046
Title: An Evaluation of Early Use of the Tortle Midliner and Intraventricular Hemorrhage (IVH) Outcomes in Premature Babies: A Randomized Controlled Trial
Brief Title: Tortle Midliner and Intraventricular Hemorrhage
Acronym: IVH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left the institution
Sponsor: Orlando Health, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB# 17.093.08
Record Dates: First submitted 2018-05-02; First posted 2018-06-01 (Actual); Results first posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Intraventricular Hemorrhage of Prematurity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Tortle Midliner (Experimental): The use of the Tortle Midliner will be in addition to the NICU department process guidelines for positioning relevant to the gestational age of the subject. The Tortle Midliner will be applied no later than 3 hours following birth under the supervision of a study investigator. The size/fit and application of the device will be according to the manufacturer's guidelines. The neutral midline head position, supine or slightly side-lying, with a bed elevation between 15° and 30° will be maintained during the first 72 hours of life.
  Interventions: Device: Tortle Midliner
- Control Group (No Intervention): All clinical care for the control group will be within NICU department process guidelines relevant to the gestational age of the subject and as ordered by physician and/or ARNP providers. The neutral midline head position with the aid of nesting and/or rolls with a bed elevation between 15° and 30° will be maintained throughout position changes during the first 72 hours of life, which is standard practice. Caregivers will document the NICU integrated flowsheet and the Sunrise electronic record with interventions regarding positioning, handling, skin assessment etc. per standard practice requirements.

INTERVENTIONS:
Device: Tortle Midliner — The Tortle Midliner will be applied in the treatment group within the first 3 hours of life and maintained until 72 hours of life.
  Arms: Tortle Midliner

SUMMARY:
The purpose of the study is to determine if early application of the Tortle Midliner for preterm infants, ≤ 3 hours following birth and with subsequent continuous use through 72 hrs. of life to ensure maintenance of optimal midline positioning (Tortle group), will impact the IVH outcome as determined by a reduction in the rate and/or severity of IVH when compared to infants receiving the standard regimen of care (Control group).

DETAILED DESCRIPTION:
Intraventricular hemorrhage (IVH) is defined as bleeding into the ventricles of the premature infant brain-the highest risk for the lowest gestational ages. IVH almost always occurs between birth and the first 72 hours of life. The four grades of IVH are based on the degree of bleeding; the greater the severity of the bleed, the more likely to have a poor outcome. Complications can include hydrocephalus, mental retardation, cerebral palsy and seizures. Neurologic sequelae can lead to death. Even for low grade bleeds the studies show the negative effects on cognitive scores and an increased incidence of learning disabilities. In addition, these same children often suffer from attention deficit disorder and other behavioral dysfunctions, which require intervention in order for the child to successfully integrate into school and society.

Since increased risk of IVH can be associated with changes of intracranial pressure, many medical protocols have established IVH bundles which are designed to help reduce fluctuations in intracranial pressure while managing the micro-preemie infant during the first few days of life.

The correlation between IVH and head positioning of the extremely low birth weight infants has made its way into research literature suggesting that venous obstruction can result from increased external pressure on the venous system when the micro-preemie infant has their head positioned to the side rather than maintaining a neutral position.

Therefore, the investigators are aiming to conduct a prospective randomized controlled trial in order to answer the research question: Does early use of the Tortle Midliner reduce the incidence and/or level of severity of intraventricular hemorrhage if used in infants born at ≤ 30 6/7 weeks and neutral position is maintained for the first 72 hours of life? The investigators hypothesize that the use of early consistent neutral positioning compared to the standard care (nested positioning) practiced in the Neonatal Intensive Care Unit (NICU) will reduce the risk of intraventricular hemorrhage in preterm infants born at ≤ 30 6/7 weeks and have a positive effect on the incidence and/or level of severity of intraventricular hemorrhage in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age less than or equal to 30 6/7 weeks at birth
2. Less than 3 hours from birth
3. Informed consent obtained from parent or legal guardian prior to reaching time point for randomization

Exclusion Criteria:

1. Presence of genetic/chromosomal abnormality, congenital hydrocephalus, congenital neuromuscular disorder, or other diagnosis determined to impact survival or generalizability of results
2. Unable to participate for any reason based on the decision of the principal investigator.
3. Infants born outside Winnie Palmer Hospital for Women and Babies

Max Age: 31 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2018-08-24 (Actual); Primary Completion 2020-01-09 (Actual); Study Completion 2020-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne C Alexander, RRT MHA DPT, Principal Investigator — Orlando Health
Locations (1):
- Orlando Health, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Study data will be shared by publication

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited in the NICU that met inclusion criteria
Pre-assignment Details: 27 subjects were randomized. 13 enrolled into the control arm and 14 in the treatment arm. 5 subjects were withdrawn after randomization ( 2 in the control arm and 3 in the treatment arm). 22 Completed study
Period: Overall Study
Arm/Group | Tortle Midliner | Control Group
Started | 14 | 13
Completed | 11 | 11
Not Completed | 3 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tortle Midliner | Control Group | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 13 | 27
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 8 | 9 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 3 | 6 | 9
  More than one race | 5 | 2 | 7
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence and Severity of Intraventricular Hemorrhage in Preterm Infants
Description: Data analysis will include descriptive statistics with means and proportions. Comparative statistics will be used to compare IVH outcomes in the two groups. IVH outcome will be determined by a reduction in the incidence and/or severity of IVH. Any additional information on data points may be described in tables and/or graphs.
Time Frame: IVH incidence and/or severity within the first week of life
Measure: Count of Participants; unit: Participants
Arm/Group | Tortle Midliner | Control Group
Number analyzed (Participants) | 11 | 11
Participants
  Incidence of IVH | 3 | 3
  Incidence of no IVH | 8 | 8

ADVERSE EVENTS:
Time Frame: Adverse events were followed from enrollment to discharge. Both groups meet criteria for a head ultrasound at 6-8 days of life. The results of the last head ultrasound and/or magnetic resonance imaging (MRI) of the brain before discharge will be collected. The duration from birth to discharge depends on the subject's medical needs. A duration of "Hospital Stay in Days" was collected as a variable. From enrollment to hospital discharge, the average timeframe was 72 days.
Description: The device, Tortle Midliner, solely impacts the skin contact areas. Only adverse events related to skin breakdown requiring wound care consultation with wound treatment will be reported as an adverse event. The principal investigator will evaluate adverse events related to skin integrity.
  Any death will be reported as a serious adverse event according to Orlando Health IRB policy.
Arm/Group | Tortle Midliner | Control Group
All-Cause Mortality (participants affected / at risk) | 0/14 | 1/13
Serious Adverse Events (participants affected / at risk) | 1/14 | 2/13
Other Adverse Events (participants affected / at risk) | 0/14 | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tortle Midliner (N=14) | Control Group (N=13)
Hypotensive shock unresponsive to aggressive vasopressor therapy (Vascular disorders) | 0 (0) | 1 (1) — Not related to device. Subject received NICU Standard of Care
Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — Subjects required increased oxygen needs and Increased work of breathing not expected in premature neonate

LIMITATIONS AND CAVEATS:
The investigator left the institution prematurely, The final study number of participants in both arms was small. More studies should be completed and evaluated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-19): https://cdn.clinicaltrials.gov/large-docs/46/NCT03543046/Prot_SAP_000.pdf